CLINICAL TRIAL: NCT00022191
Title: Randomized Phase III Study Comparing Paclitaxel/Cisplatin/Gemcitabine and Cisplatin/Gemcitabine in Patients With Metastatic or Locally Advanced Urothelial Cancer Without Prior Systemic Therapy
Brief Title: Cisplatin Plus Gemcitabine With or Without Paclitaxel in Treating Patients With Stage IV Urinary Tract Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Groupe D'Etude des Tumeurs Uro-Genitales (Other); Institute of Cancer Research, United Kingdom (Other); Central European Cooperative Oncology Group (Other); NCIC Clinical Trials Group (Network); SWOG Cancer Research Network (Network); German Association of Urologic Oncology (Other); Spanish Oncology Genito-Urinary Group (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30987; EORTC-30987; CAN-NCIC-BL7; CECOG-EORTC-30987; GAUO-EORTC-30987; GETUG-EORTC-30987; SOGUG-EORTC-30987; SWOG-30987; NCRI-CRUK-BA11; MRC-BA11
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage IV bladder cancer; transitional cell carcinoma of the bladder; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Cisplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective for urinary tract cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin plus gemcitabine with or without paclitaxel in treating patients who have stage IV urinary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the duration of survival of patients with stage IV transitional cell carcinoma of the urothelium treated with cisplatin and gemcitabine with or without paclitaxel.
* Compare the duration of progression-free survival, response rates, and duration of response in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, WHO performance status (0 vs 1), and presence of metastatic disease (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 1 hour on day 1 or 2. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive paclitaxel IV over 1 hour on days 1 and 8 followed by cisplatin IV over 1 hour on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for at least 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 610 patients (305 per treatment arm) will be accrued for this study within 3.04 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV transitional cell carcinoma of the urothelium (pure or mixed) including bladder, urethra, ureter, and renal pelvis

  * T4b, any N OR any T, N2-3 OR M1
* Ineligible for surgery or radiotherapy with curative intent
* Measurable or evaluable disease
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.25 times normal
* AST or ALT less than 2.5 times normal

Renal:

* Glomerular filtration rate at least 60 mL/min
* Calcium normal or clinically insignificant

Cardiovascular:

* No clinically significant cardiac arrhythmia
* No congestive heart failure
* No complete bundle branch block
* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No grade 3 or 4 infection without neutropenia
* No other serious concurrent systemic disorder that would preclude study therapy
* No mental disorder that would preclude study compliance
* No grade II or greater neuropathy
* No other prior or concurrent malignancy except appropriately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, or incidental prostate cancer (T1, Gleason score no greater than 6, and PSA less than 0.5 ng/mL)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior investigational biologic agents (e.g., antiangiogenic products, signal transduction pathway inhibitors, immunomodulators, or monoclonal antibody therapy)
* At least 4 weeks since prior immunotherapy

Chemotherapy:

* No prior systemic chemotherapy
* At least 4 weeks since prior local intravesical chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No more than 1 prior course of radiotherapy
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* Prior urological procedures to relieve urinary tract obstruction and improve renal function allowed (e.g., ureteral stent or percutaneous nephrostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2001-05; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD, PhD, Study Chair — Vall d'Hebron University Hospital; Stephane Culine, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle; Michael Leahy, MBChB, FRACP, FRCP, FRC Path, Study Chair — Fremantle Hospital; Christoph Zielinski, MD, Study Chair — Allgemeines Krankenhaus - Universitatskliniken; Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada; David C. Smith, MD, Study Chair — University of Michigan Rogel Cancer Center; Andreas Boehle, MD, Study Chair — Universitaetsklinikum Schleswig-Holstein - Campus Luebeck; Jose Baselga, MD, Study Chair — Vall d'Hebron University Hospital
Locations (234):
- United States (58):
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Del Rio, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Southwest Cancer and Research Center at University Medical Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
- Fremantle Hospital, Fremantle, Western Australia, Australia
- Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
- Canada (69):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic at Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Providence Health Care - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre - Sudbury, Greater Sudbury, Ontario
  - Hamilton and District Urology Association, Hamilton, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchner, Ontario
  - London Health Sciences Centre, London, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, North York, Ontario
  - Male Health Centre - Oakville, Oakville, Ontario
  - Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma Reginal Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Male Health Centre - North York, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Prince Edward Island Cancer Center at Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Complexe Hospitalier de la Sagamie, Chicoutimi, Quebec
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Québec, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Denmark (2):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (24):
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Hopital Lapeyronie-CHU Montpellier, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Tenon, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Medico-Chirurgical Foch, Suresnes
  - Centre Antoine Lacassagne, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (34):
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - Charite Humboldt - University Berlin, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Helios - Klinik Blankenhain, Blankenhain
  - Universitaetsklinikum Bonn, Bonn
  - Staedtische Kliniken Dortmund, Dortmund
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - St. Markus Krankenhaus, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Fulda, Fulda
  - Martin Luther Universitaet, Halle
  - Marienkrankenhaus, Hamburg
  - Universitat des Saarlandes Innere Medizin 1, Hamburg
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Staedtisches Krankenhaus Sued, Lübeck
  - Medizinische Universitaet Luebeck, Lübeck
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Klinikum der Stadt Mannheim, Mannheim
  - University of Marburg, Marburg
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Kinderheilkunde, Münster
  - Klinikum Neubrandenburg, Neubrandenburg
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Paracelsus Karankenhaus Ruit, Ostfildern
  - Asklepios Klinik Pasewalk, Pasewalk
  - Diakonie - Krankenhaus, Rotenburg (Wümme)
  - Johanniter Kankenhaus Stendal, Stendal
  - Katharinenhospital, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaet Ulm, Ulm
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Klinikum St. Marien, Wuppertal
  - Witten University - Klinikum Wuppertal, Wuppertal
- National Institute of Oncology, Budapest, Hungary
- Israel (2):
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (2):
  - Ospedale Santa Croce, Cuneo
  - Istituto Scientifico H.San Raffaele, Milan
- Netherlands (5):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Jeroen Bosch Ziekenhuis, NL'S Hertogenbosch
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
  - University Hospital - Rotterdam Dijkzigt, Utrecht
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (20):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Arquitecto Marcide, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario De Guadalajara, Guadalajara
  - Hospital Cuidad de Jaen, Jaén
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario - Malaga, Málaga
  - Hospital Son Dureta, Palma de Mallorca
  - Hospsital de Sabadell, Sabadell
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Consorci Sanitari De Terrassa, Terrassa
  - Instituto Valenciano De Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Rio Hortega, Valladolid
  - Hospital General De Vic, Vic
  - Hospital Clinico Universitario, Zaragoza
- United Kingdom (8):
  - Princess Royal Hospital, Hull, England
  - St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals NHS Trust, London, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Marsden Hospital - Sutton, Sutton, England
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales

REFERENCES:
- [Result] Bellmunt J, von der Maase H, Mead GM, et al.: Randomized phase III study comparing paclitaxel/cisplatin/gemcitabine (PCG) and gemcitabine/cisplatin (GC) in patients with locally advanced (LA) or metastatic (M) urothelial cancer without prior systemic therapy: EORTC30987/Intergroup study. [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA5030, 242s, 2007.